CLINICAL TRIAL: NCT00962728
Title: Assessment of Inspiratory Breathing Devices to Improve Orthostatic Tolerance in Postural Orthostatic Tachycardia Syndrome
Brief Title: Breathing Device in Postural Orthostatic Tachycardia Syndrome (POTS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alfredo Gamboa (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Alfredo Gamboa, Research Assistant Professor of Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 090609
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Postural Tachycardia Syndrome; Postural Orthostatic Tachycardia Syndrome
Keywords: heart rate; tachycardia; orthostatic intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Tachycardia; Orthostatic Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITD breathing device (Experimental): Breathing through the Res-Q-Gard ITD device from Advanced Circulatory Systems Inc.
  Interventions: Device: Inspiratory Threshold Device (Res-Q-Gard ITD)
- Sham Device (Sham Comparator): Breathing through a respiratory particulate filter (Model 002850P, Sims Portex Inc, Keene NH) which will have minimal resistance.
  Interventions: Device: Sham Inspiratory Threshold Device

INTERVENTIONS:
Device: Inspiratory Threshold Device (Res-Q-Gard ITD) — Patient will breathe through this device attached to a mouthpiece during assessment of orthostatic tolerance.
  Other Names: Res-Q-Gard ITD device 7.0 (Ref:12-0463-000)
  Arms: ITD breathing device
Device: Sham Inspiratory Threshold Device — Breathing through a respiratory particulate filter (Model 002850P, Sims Portex Inc, Keene NH) which will have minimal resistance.
  Other Names: Model 002850P, Sims Portex Inc, Keene NH
  Arms: Sham Device

SUMMARY:
The investigators will test whether breathing through an inspiratory resistance device will improve the ability to be upright and decrease heart rate increases on standing in patients with postural tachycardia syndrome.

DETAILED DESCRIPTION:
Chronic orthostatic intolerance, sometimes known as the postural tachycardia syndrome (POTS), is the most common disorder among patients seen at several centers specializing in diseases of the autonomic nervous system. It affects an estimated 500,000 people in the United States alone. POTS (excessive increase in heart rate [>30 min-1] on standing associated with orthostatic symptoms [including palpitation, chest pain syndrome, dyspnea on standing, mental clouding and difficulties with concentration], in the absence of orthostatic hypotension) can produce substantial disability among otherwise healthy people. Patients with POTS typically feel tired and run down. Many also report a myriad of symptoms that are hard to categorize, often involving fatigue. One study, from the Mayo Clinic, found that patients with POTS had a diminished quality of life when measured using a standard health status instrument (SF-36).

In this pilot study, we will test the hypothesis that breathing through an inspiratory resistance device will improve orthostatic tolerance and reduce orthostatic tachycardia in patients with postural tachycardia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center
* Increase in heart rate ≥ 30 beats/min with position change from supine to standing (10 minutes)
* Chronic symptoms consistent with POTS that are worse when upright and get better with recumbence
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Inability to give, or withdrawal of, informed consent
* Pregnant
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Magnitude of orthostatic heart rate increase on upright posture | 10 min

SECONDARY OUTCOMES:
Symptoms rating with upright posture | 10 min
Hemodynamic changes on upright posture | 10 min

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Convertino VA, Ryan KL, Rickards CA, Cooke WH, Idris AH, Metzger A, Holcomb JB, Adams BD, Lurie KG. Inspiratory resistance maintains arterial pressure during central hypovolemia: implications for treatment of patients with severe hemorrhage. Crit Care Med. 2007 Apr;35(4):1145-52. doi: 10.1097/01.CCM.0000259464.83188.2C. PMID 17334239
- [Background] Convertino VA, Ratliff DA, Crissey J, Doerr DF, Idris AH, Lurie KG. Effects of inspiratory impedance on hemodynamic responses to a squat-stand test in human volunteers: implications for treatment of orthostatic hypotension. Eur J Appl Physiol. 2005 Jul;94(4):392-9. doi: 10.1007/s00421-005-1344-1. Epub 2005 Apr 28. PMID 15864634
- [Derived] Gamboa A, Paranjape SY, Black BK, Arnold AC, Figueroa R, Okamoto LE, Nwazue VC, Diedrich A, Plummer WD, Dupont WD, Robertson D, Raj SR. Inspiratory resistance improves postural tachycardia: a randomized study. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):651-8. doi: 10.1161/CIRCEP.114.002605. Epub 2015 Mar 19. PMID 25792354
- See also: Vanderbilt Autonomic Dysfunction Center — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction